CLINICAL TRIAL: NCT03016364
Title: Application Software in Dosage Adjustment for Advanced Cancer Patients With Pain
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Peng Liu, Attending Physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFH2016-3-4025
Record Dates: First submitted 2017-01-09; First posted 2017-01-10 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Pain; Physicians; Oxycodone
MeSH Terms: conditions — Pain

ARMS (1):
- APP in dosage adjustment (Experimental): Through the guidance of APP software, clinical doctors try to adjust the dose of Oxycodone Hydrochloride Prolonged-release Tablets for advanced patient's with cancer pain.
  Interventions: Device: APP software

INTERVENTIONS:
Device: APP software — A software used to by physicians to adjust the dose of Oxycodone Hydrochloride Prolonged-release Tablets for advanced patient's with cancer pain

SUMMARY:
The purpose of this trial is to determine whether Application (APP) would help clinical doctors to adjust the dose of Oxycodone Hydrochloride Prolonged-release Tablets in advanced patients with cancer pain.

ELIGIBILITY:
Inclusion Criteria:

* a histologically confirmed diagnosis of Cancer or Sarcoma
* advanced patients with severe cancer pain(score >3)
* having used or expected to use the Oxycodone Hydrochloride Prolonged-release Tablets

Exclusion Criteria:

* allergic to Oxycodone Hydrochloride Prolonged-release Tablets, or other reasons (determined by clinical doctors) unable to use the Opioids

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | upto 8 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China